CLINICAL TRIAL: NCT01356264
Title: Multimodal Prehabilitation to Enhance Functional Recovery After Colorectal Surgery: a Randomized Controlled Trial
Brief Title: Multimodal Prehabilitation for Colorectal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Society of American Gastrointestinal and Endoscopic Surgeons (Other); Immunotec Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Liane S. Feldman, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEN# 11-004
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer; Colorectal Cancer Stage III
Keywords: colorectal cancer; colorectal surgery; prehabilitation; surgical recovery; exercise; referred for scheduled resection
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- multimodal prehabilitation begun preop (Experimental): The prehabilitation program will begin several weeks preop and continue in the postoperative period
  Interventions: Behavioral: multimodal prehabilitation
- Multimodal prehabilitation begun postop (Active Comparator): The prehabilitation program will begin after the surgery.
  Interventions: Behavioral: multimodal prehabilitation

INTERVENTIONS:
Behavioral: multimodal prehabilitation — multimodal prehabilitation program based on exercise, supplemental nutrition and psychological support starting 3-5 weeks before surgery and continuing postoperative for up to 8 weeks
  Arms: multimodal prehabilitation begun preop
Behavioral: multimodal prehabilitation — multimodal prehabilitation program based on exercise, supplemental nutrition and psychological support beginning postoperative and continuing for up to 8 weeks
  Arms: Multimodal prehabilitation begun postop

SUMMARY:
Despite advances in surgical care, the incidence of postoperative complications and prolonged recovery following colorectal surgery remains high. Efforts to improve the recovery process have primarily focused on the intraoperative (eg, minimally invasive surgery, afferent neural blockade) and post-operative periods (eg, "fast track" early nutrition and mobilization. The pre-operative period may in fact be a better time to intervene in the factors that contribute to recovery. The process of enhancing functional capacity of the individual in anticipation of an upcoming stressor has been termed "prehabilitation". Based on the notion that preoperative exercise would have an impact on recovery of functional capacity after colorectal surgery, our group recently conducted a randomized controlled trial. Subgroup analysis identified that patients whose functional exercise capacity improved preoperatively, regardless of exercise technique, recovered well in the postoperative period. However, one-third of patients deteriorated preoperatively despite the exercise regimen, and these patients were also at greater risk for prolonged recovery after surgery. These results suggested that exercise alone is not sufficient to attenuate the stress response in all patients. In the present trial, the impact of a multimodal prehabilitation intervention composed of exercise, nutritional supplement and psychological well-being begun in the preoperative period will be compared to one begun in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* referred for scheduled surgery for nonmetastasized colorectal cancer
* age > 18 years old

Exclusion Criteria:

* asa 4-5
* Poor English or French comprehension
* severe co-morbid disease interfering with ability to perform exercise at home or complete testing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
six minute walk test | baseline, preop, 4 weeks, 8weeks postop
  6 MWT is a patient-relevant measure of functional walking capacity, reflective of the activities of daily living. Subjects are instructed to walk back and forth, in a 20 m stretch of hallway, for six minutes, at a pace that would make them tired by the end of the walk. The distance in meters is recorded. Reference equations are available for calculating percent of age- and gender-specific norms.

SECONDARY OUTCOMES:
Health-related quality of life | baseline, preop, 4 weeks, 8 weeks
  The SF-36 is the most widely used HRQL measure and has been validated for surgical population; Canadian norms are also available. It incorporates behavioural functioning, subjective well-being and perceptions of health by assessing, on a 0 to 100 scale, eight health concepts.
physical activity level | baseline, preop, 4 weeks, 8 weeks
  Physical activity level will be measured through the Community Health Activities Model Program for Seniors (CHAMPS) questionnaire. CHAMPS is a self-reported measure of physical activity, comprising 41 activities evaluated according to the total number of hours done during an average week. Each physical activity is assigned a MET (metabolic equivalent) value yielding average weekly caloric expenditure for the listed physical activities
Depression and anxiety | baseline, preop, 4 weeks, 8 weeks
  Depression and anxiety will be assessed by The Hospital Anxiety and Depression Scale (HADS), a 14-question measure with seven items each for depression and anxiety. HADS generates separate scores for anxiety and depression as well as a combined score of psychological distress.
nutritional status | baseline, preop, 4 weeks, 8 weeks
  Nutritional status will be assessed at baseline by measuring body mass index (BMI), body weight loss over the preceding three months (> 10% ), and/or serum albumin < 35 g -1 will define poor nutritional status.
postoperative complications | 4 weeks
  Classified by Clavien Scale
Fatigue | baseline, preop, 4 wks, 8 wks
  Fatugue Index

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub3. PMID 37162250
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252
- [Derived] Gillis C, Fenton TR, Sajobi TT, Minnella EM, Awasthi R, Loiselle SE, Liberman AS, Stein B, Charlebois P, Carli F. Trimodal prehabilitation for colorectal surgery attenuates post-surgical losses in lean body mass: A pooled analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1053-1060. doi: 10.1016/j.clnu.2018.06.982. Epub 2018 Jul 9. PMID 30025745
- [Derived] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535